CLINICAL TRIAL: NCT04105556
Title: The Effect of Nursing Care Based on Kolcaba's Comfort Theory to the Comfort and Components of the Child and Parents Who Are Planned for Male Circumcision Operation
Brief Title: Male Circumcision and Comfort Theory
Acronym: Comfort Theory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Fahriye Celik, Research Assistant, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SuleymanDUnursingcare
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Nursing Caries
Keywords: Male Child; Comfort Theory; Fear; Male Circimcision; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Type of intervention, testing the comfort and components of children and parents of the circumcision operation plan with Nursing Care Based on Kolcaba's Comfort Theory
Who Masked: Participant, Care Provider
Masking Description: Male child and care provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nursing Care Based on Kolcaba's Comfort Theory (Experimental): In this study, nursing care based on Kolcaba's Comfort Theory, which continues throughout the perioperative period, was applied to children and their parents.
  Care was given when the child and his / her parents applied to the outpatient clinic for anesthesia consultation on the working day before the operation, and care was continued in the day surgery unit. On the 1st and 3rd days after discharge, the researcher provided tele-monitoring and consultancy services. In addition, communication with the parents was maintained at all times as needed. Care was terminated on the 10th day after discharge. The time of the study was approximately 12-14 days for each child and his / her parents.
  Nursing care consists of 3 types of comfort-oriented care interventions. These interventions;
  1. Standard maintenance interventions,
  2. Emotional focused comfort care interventions,
  3. Cognitive and functional comfort care interventions.
  Interventions: Other: Nursing Care Based on Kolcaba's Comfort Theory
- Routine hospital schedule (No Intervention): The researcher sincerely answered all questions asked by the control group during the perioperative period.
  After the post-discharge post-tests, the control group was given a gift of medal of courage, a story book and a training booklet prepared for the parents after the policlinic control on the 10th postoperative day, and the training was given to the intervention group.

INTERVENTIONS:
Other: Nursing Care Based on Kolcaba's Comfort Theory — In this study, nursing care based on Kolcaba's Comfort Theory, which continues throughout the perioperative period, was applied to children and their parents.
  Other Names: • Pre-surgical preparation program • Comfort-oriented care • Tele-monitoring and consultancy
  Arms: Nursing Care Based on Kolcaba's Comfort Theory

SUMMARY:
Aim: Male circumcision is one of the oldest and most commonly performed surgical procedures in the world and in our country. Circumcision, which concerns such a large population, is a stressful, traumatic, negative experience. Impairment in comfort is a condition in which a child who is scheduled for circumcision operation often suffers. Physical, emotional, sociocultural and environmental factors contribute to the formation of this condition. Comfort Theory is a nursing model that makes it easier for the caregivers to see their problems more systematically and to plan more easily. In the literature review, no studies have been found to determine the effect of nursing care based on Kolcaba Konfors Comfort Theory to the comfort and components of the children and their parents who have undergone circumcision operation. Therefore, this study was needed. In this study, nursing care based on Kolcaba's Comfort Theory, which continues throughout the perioperative period, was applied to children and their parents.

Method: In this study, the effect of nursing care based on Kolcaba's Comfort Theory on fear, anxiety, pain, comfort and anxiety in parents and health care satisfaction was tested in children. Care was given when the child and his / her parents applied to the outpatient clinic for anesthesia consultation on the working day before the operation, and care was continued in the day surgery unit. On the 1st and 3rd days after discharge, the researcher provided tele-monitoring and consultancy services. In addition, communication with the parents was maintained at all times as needed. Care was terminated on the 10th day after discharge. The time of the study was approximately 12-14 days for each child and his / her parents.

The sample of the study was determined as 120 boys and their parents (60 control each, 60 intervention each). In this study, standard nursing care will be applied to the control group and nursing care based on Kolcaba's Comfort Theory will be applied to the intervention group. The data will be collected with the Child and Family Descriptive, VAS, Children's State Anxiety (CSA) and Children's Fear Scale (CFS), Comfort Behavior Checklist, Spielberger State Anxiety Scale, PedsQL Health Care Satisfaction Scale.

DETAILED DESCRIPTION:
In this study, nursing care based on Kolcaba's Comfort Theory, which continues throughout the perioperative period, was applied to children and their parents.

Care was given when the child and his / her parents applied to the outpatient clinic for anesthesia consultation on the working day before the operation, and care was continued in the day surgery unit. On the 1st and 3rd days after discharge, the researcher provided tele-monitoring and consultancy services. In addition, communication with the parents was maintained at all times as needed. Care was terminated on the 10th day after discharge. The time of the study was approximately 12-14 days for each child and his / her parents.

Nursing care consists of 3 types of comfort-oriented care interventions. These interventions;

1. Standard maintenance interventions,
2. Emotional focused comfort care interventions,
3. Cognitive and functional comfort care interventions.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 4-7
* No previous surgical experience of the child
* Lack of chronic disease, disability and developmental delay of the child
* The child or his / her parent does not have a special situation that causes difficulties in understanding and perception.
* Parent's ability to read and write in Turkish

Exclusion Criteria:

* Child / parent who does not volunteer to participate in the study
* Children who are not cared for at least two relatives during the surgical procedure

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male circumcision
Enrollment: 120 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Comfort Behaviors Checklist | In two weeks
  Comfort Behaviors Checklist was developed in 1989 by Kolcaba. Developed as a last resort, data collectors are used to rate a patient's apparent comfort. While not as desirable as actually asking a patient about his or her comfort, the instrument can fill a gap regarding data collection in comatose, very frail (as in terminal), or cognitively limited patients. Kolcaba and DiMarco (2005) reported that postoperative comfort in children can be assessed using the Comfort Behavior Checklist. The reliability and validity study of our country was conducted by Unutkan and Balcı Yangın (2018).
VAS | In two weeks
  The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. Instructions, time period for reporting, and verbal descriptor anchors have varied widely in the literatüre. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]). Varies, but most commonly respondents are asked to report "current" pain intensity or pain intensity "in the last 24 hours." A higher score indicates greater pain intensity. Based on the distribution of pain VAS scores in postsurgical patients who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain VAS have been recommended: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm)
Children's Fear Scale | In two weeks
  It was developed by McMurty et al. (2011). The validity and reliability study of the Turkish Children's Fear Scale was conducted by Özalp Gerçeker and colleagues in 2017. The scale can be used to assess fear in children aged 4-10 years. The CFS consists of five drawn facial expressions ranging from neutral expression (0 = no anxiety) to the frightened face (4 = severe anxiety), and can be easily evaluated by parents, researchers, and healthcare professionals who care for the child. It is a scale of one item. CFS was developed based on the Faces Anxiety Scale developed to measure the anxiety or fear of adults in the intensive care unit of McKinley et al. (2003).
Children's Anxiety Meter-State (CAM-S) | In two weeks
  The scale was developed by Ersig et al. (2013). The Turkish validity and reliability study of the scale was conducted by Özalp Gerçeker et al. The scale can be used to assess anxiety in children aged 4-10 years. The score can vary from 0 to 10 (Ersig et al., 2013)
The State-Trait Anxiety Inventory (STAI) | In two weeks
  In the study, STAI will be used to determine the anxiety of parents. It was developed by Spielberger et al. (1970). The Turkish validity and reliability study of the STAI was conducted by Öner and Le Compte in 1983. The scale is a 4-point Likert type and contains two 20-item expressions. Direct expressions express negative emotions and reversed expressions express positive emotions. It was reported that the Cronbach Alpha internal consistency coefficient ranged between α = 0.83 and 0.87 (Sarıtaş and Büyükbayram, 2016).
The PedsQL (Pediatric Quality of Life InventoryTM) | In two weeks
  The PedsQL will be used to measure the level of health care satisfaction of parents. The scale consists of 25 questions. The questions in the scale are aimed at measuring satisfaction with medical care services and psychosocial satisfaction. Cronbach Alpha internal consistency coefficient of the scale, which was validated by Varni (1999), was found to be α = .96. Scale was adapted to Turkish by Ulus and Kublay (2012).

CONTACTS AND LOCATIONS:
Overall Officials: Emine EFE, Study Director — Akdeniz Universty
Locations (1):
- Fahriye PAZARCIKCI, Isparta, Türki̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagner D, Byrne M, Kolcaba K. Effects of comfort warming on preoperative patients. AORN J. 2006 Sep;84(3):427-48. doi: 10.1016/s0001-2092(06)63920-3. PMID 17004666
- [Background] Dowd T, Kolcaba K, Steiner R, Fashinpaur D. Comparison of a healing touch, coaching, and a combined intervention on comfort and stress in younger college students. Holist Nurs Pract. 2007 Jul-Aug;21(4):194-202. doi: 10.1097/01.HNP.0000280931.75883.ae. PMID 17627198
- [Background] Dowd T, Kolcaba K. Two interventions to relieve stress in college students. Beginnings. 2007 Winter;27(1):10-1. No abstract available. PMID 17381027
- [Background] Kolcaba K, Tilton C, Drouin C. Comfort Theory: a unifying framework to enhance the practice environment. J Nurs Adm. 2006 Nov;36(11):538-44. doi: 10.1097/00005110-200611000-00010. PMID 17099440
- [Result] Kolcaba K, DiMarco MA. Comfort Theory and its application to pediatric nursing. Pediatr Nurs. 2005 May-Jun;31(3):187-94. PMID 16060582